CLINICAL TRIAL: NCT01989832
Title: Pharmaco-economical Study in Kidney Transplantation
Acronym: EPHEGREN
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10007
Record Dates: First submitted 2013-11-04; First posted 2013-11-21 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2014-06

CONDITIONS: Renal Transplant
Keywords: cohort; pharmaco-economic; kidney; transplantation; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biological and clinical Data collected

SUMMARY:
The prevalence of renal acute rejection in transplantation is reduced thanks to the optimized use of immunosuppressive drugs. However, graft survival at ten years has not improved since then; this may be explained in part by the toxicity of these drugs, viral infections, and other comorbidities (diabetes, cardiovascular diseases …).

According to transplant center, strategies for the combination of immunosuppressive drugs are different, and probably involve a difference in the global cost of patient management. There is no recommendation in France to establish similar practices.

EPHEGREN is an observational, prospective, multicentric, pharmacoeconomic study for the renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the first month of renal graft, or patients already included in an other epidemiological French study (EPIGREN) in the 0-6 month period
* Men of women aged more than 18 years
* Patients able to exercise in writing their informed and free consent to participate to the biological collection
* Patients not opposing to collect their medical data
* Patients registered with a social security system
* Patients able to complete the questionnaires

Exclusion Criteria:

* Patients aged less than 18 years and patients under guardianship
* Patients with a follow-up at another center other than those part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: renal transplant patients
Sampling Method: Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of Death | 4 years

SECONDARY OUTCOMES:
to examine nature, dose and exposure in immunosuppresseurs. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges, France